CLINICAL TRIAL: NCT01361451
Title: Myotrace: A Phase II Evaluation of a Novel Critical Illness Monitoring System
Brief Title: Myotrace: An Evaluation of a Novel Critical Illness Monitoring System
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RJ111/N002
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2010-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: parasternal electromyogram; neural respiratory drive; chronic obstructive pulmonary disease; respiratory physiology; Acute exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — It is envisaged that a subset of patients will have venous blood samples taken for future analysis for inflammatory cytokines
Oversight: Data Monitoring Committee: No

SUMMARY:
There are 24,000 admissions each year to Intensive Care Units (ICU) in the United Kingdom due to pneumonia, asthma and a common condition called chronic obstructive pulmonary disease (COPD), with rates of death of 10%, 40% and 50%, respectively. These conditions account for 10% of all ICU admissions. It is therefore important to find out if it would be possible to detect deteriorations in patients with breathing problems early, in order to increase appropriately their level of care.

Clinical early warning scores (EWS) are used in many hospitals to detect patients whose medical condition is getting worse, and who are likely to need admission to intensive care or high dependency care units. EWS are usually calculated from several measurements taken from the patient, such as blood pressure, temperature and heart rate. However, they are often inaccurate as they need to be calculated manually by nursing staff from a number of measurements taken from a variety of different devices. Furthermore, even when accurately calculated, it is not clear how helpful EWS are in predicting whether or not patients will deteriorate.

Neural respiratory drive (NRD) is an objective indicator of breathlessness, and can be derived from the amount of electrical activity occurring in certain muscles used in breathing. The Myotrace system measures this electrical activity, as well as measurements such as rate of breathing and heart rate. It then analyses these measurements together to help identify patients at risk of deterioration.

This study will use Myotrace to monitor patients with severe breathing difficulties due to an acute worsening of chronic obstructive pulmonary disease, for early identification of failure to respond to medical treatment.

Patients will be recruited at St. Thomas' Hospital.

This research is funded by the Guy's and St. Thomas' Charity.

DETAILED DESCRIPTION:
Admissions to hospital due to breathing difficulties are common. When these patients' medical condition worsens, the deterioration is often not noticed until the patient needs to be moved to an area of the hospital that provides higher levels of care, e.g. intensive care unit or high-dependency unit.

Early warning scores (EWS) have been designed to help medical and nursing staff identify patients at risk of deteriorating. These scores are usually calculated from patient measurements such as blood pressure and heart rate. It is not clear how effective these scores are in preventing patient deterioration, or the need for intensive or high-dependency care. The investigators therefore need another means of identifying patients at risk of deterioration, particularly in those with breathing difficulties.

Neural respiratory drive is a term used to describe the nervous system's response to the need for increased breathing, and may be helpful in predicting whether patients admitted to hospital with breathing difficulties will deteriorate. This response may be measured as the amount of electrical activity that occurs in the muscles associated with breathing, which are supplied with nerves that deliver electrical messages to the fibres that make up muscle.

The main breathing muscle in the body is the diaphragm, a sheet of muscle lying beneath the lungs, which, when it contracts, moves downwards and draws air into the lungs. Although the electrical activity in the diaphragm may be measured, this can only be achieved using a technique that involves passing an electrical probe into a patient's oesophagus, or gullet. This is not easy to do in a patient that has been admitted unwell to hospital with breathing difficulties.

Therefore, a technique has been developed to measure the electrical activity that occurs in the parasternal muscles. These muscles lie either side of the sternum, or breast bone, and are particularly important breathing muscles in patients with chronic obstructive pulmonary disease (COPD), a lung disease commonly associated with smoking. Parasternal muscle electrical activity can be measured from probes attached to the skin of the chest wall, and can therefore be achieved more easily than measuring diaphragm electrical activity.

Previous studies have shown that parasternal electrical activity is comparable to diaphragm electrical activity in patients with COPD, and is a useful measure of neural respiratory drive in patients with COPD. Neural respiratory drive has been shown to be increased in patients with stable COPD.

A pilot study involving 25 patients with COPD showed that daily measurements of parasternal electrical activity are possible in patients admitted to hospital with acute worsening of COPD. This study also demonstrated that the amount of parasternal electrical activity reflected the degree of breathlessness experienced by patients with acute worsening of COPD. Importantly, this study showed that measures related to parasternal electrical activity, and hence neural respiratory drive, were significantly different in patients whose medical condition deteriorated, compared with those that improved with treatment. Clinical early warning scores were not significantly different between these two groups. Furthermore, measures related to parasternal electrical activity were able to predict whether a patient with an acute worsening of COPD would be readmitted to hospital within 7 and 14 days of discharge.

Therefore, measurement of parasternal activity may be helpful in predicting deterioration due to treatment failure in patients admitted to hospital with acute worsening of COPD. However, as the pilot study was performed on a small number of patients, a larger clinical trial of the Myotrace system, which acquires, processes and analyses this information, is needed to demonstrate this conclusively. This is the purpose of the current study.

Patients with acute worsening of COPD, as diagnosed by a doctor, will be recruited from the Emergency Department or the acute admissions wards at St. Thomas' Hospital, London. On admission, it is normal practice for the Patient At Risk (PAR) score to be recorded. This is the Early Warning Score used at Guy's and St. Thomas' NHS Foundation Trust (GSTFT).

Patients will usually have had a blood test to check blood gas content as part of their normal medical care.

The research team will identify potential candidates for the study in two ways: firstly, directly from the Emergency Department; secondly, following admission, when new patients with COPD will have been seen by the medical team directly responsible for the patient's medical care or COPD outreach team. The research team will liaise with the medical and COPD outreach teams to identify potential participants.

Potential candidates then be given oral and written information about the study. Patients' capacity to consent will be assessed at this time. Patients will be given the opportunity to consider participating in the study for 3 hours, after which written consent will be sought. The relatively short period of time for consideration is due to the potential for patients' medical condition to change rapidly.

Following recruitment, patients will be asked about the history of their breathing difficulties. Height and weight will be recorded where possible. Patients will be asked how breathless they normally feel when stable (MRC dyspnoea score) and how breathless they currently feel (visual-analogue scale).

A further blood sample may be taken to assess for markers of inflammation on enrollment; inflammation in COPD remains poorly understood, and it is intended that these blood tests will inform further studies into this process.

Parasternal electromyogram (EMG) electrodes will then be attached to the patient's chest, either side of the sternum (breast bone), to measure muscle electrical activity, breathing rate and heart rate, using the Myotrace system. Electrode position will be marked with indelible ink, to make sure that electrodes are re-attached to the chest wall in the same place after washing or other activities. Electrodes will also be applied to the neck and the abdomen, as muscles in these areas also contribute significantly to breathing.

The patient will first be asked to sniff as hard as possible through the nose, to measure the maximum electrical activity that the parasternal muscles can generate. All other measures of muscle electrical activity will then be expressed as a percentage of this maximum.

Parasternal muscle electrical activity, breathing rate and heart rate will be measured using the Myotrace system, as well as normal bedside measurements of temperature, blood pressure and oxygen levels. An Early Warning Score will also be calculated (the PAR score). Measurements will be taken for 20 minutes three times a day (at around 9am, 12 noon and 6pm), until the patient is discharged from hospital.

Patients will also wear an activity monitor, either on the wrist or around the neck. This will monitor the patient's physical activity, which is known to be related to decline in breathing function in patients with COPD. The patient will be asked to keep the monitor on throughout their hospital stay and for up to three months after discharge. The activity monitors are very light to wear and very well-tolerated by patients.

Patients will be asked to complete a diary card recording their symptoms three times a day during Myotrace measurements. Tests of breathing function (spirometry) will also be performed.

The research team will not inform the medical team looking after the patient of the results of the tests, whilst the patient remains in hospital. When the patient is ready to be discharged home, he/she will be asked to complete a number of questionnaires about their breathing difficulties and their quality of life. A further blood sample will be taken at this stage for markers of inflammation.

The research team will note whether the patient has been discharged with support from the COPD outreach, to see whether there is any relationship between being offered supported discharge and muscle electrical activity.

Patients will be offered follow-up appointments with the research team at St. Thomas' Hospital one month and three months after discharge from hospital. During this appointment, further blood tests may be taken to check for blood gas content and any persisting infection or inflammation. The patient will be asked to complete further questionnaires relating to breathlessness and quality of life. Measurements of breathing muscle electrical activity will be repeated, and patients' physical activity data analysed.

ELIGIBILITY:
Inclusion Criteria:

* Admitted patients with physician diagnosis of AECOPD
* Smoking history ≥ 10 pack years, consistent with COPD
* Expected to remain an inpatient for ≥ 24 hours
* Age ≥ 35 years
* Able to give informed consent to participation in the study

Exclusion Criteria:

* Requirement for immediate mechanical ventilation at admission
* Presence of another acute pathology (such as pulmonary embolism, pneumonia or pulmonary oedema) to explain the acute presentation
* Presence of other severe medical problem, e.g. cancer
* Psychological and social factors that would impair compliance with the study schedule

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalised patients with acute exacerbation of chronic obstructive pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Readmission to hospital | 28 days
  Readmission to hospital within 28 days of discharge, following acute exacerbation of COPD

SECONDARY OUTCOMES:
Length of hospital stay | expected to be 2-9 days
Physical activity | Up to 3 months after discharge from hospital
  as measured by two types of activity monitor during hospital stay and up to 3 months after discharge
Treatment failure | up to 1 month following admission
  * Transfer to High Dependency Unit
  * Arterial blood gas demonstrating respiratory failure requiring non-invasive ventilation, if appropriate
  * Transfer to ICU
  * Arterial blood gas demonstrating respiratory failure requiring invasive ventilation, if appropriate
  * Hospital Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Hart, PhD, Study Director — Guy's and St Thomas' NHS Foundation Trust; Eui-Sik Suh, MBBS, Principal Investigator — King's College London
Locations (1):
- St. Thomas' Hospital, London, United Kingdom

REFERENCES:
- [Derived] Patout M, Meira L, D'Cruz R, Lhuillier E, Kaltsakas G, Arbane G, Suh ES, Hart N, Murphy PB. Neural respiratory drive predicts long-term outcome following admission for exacerbation of COPD: a post hoc analysis. Thorax. 2019 Sep;74(9):910-913. doi: 10.1136/thoraxjnl-2018-212074. Epub 2019 Apr 26. PMID 31028235
- [Derived] Suh ES, Mandal S, Harding R, Ramsay M, Kamalanathan M, Henderson K, O'Kane K, Douiri A, Hopkinson NS, Polkey MI, Rafferty G, Murphy PB, Moxham J, Hart N. Neural respiratory drive predicts clinical deterioration and safe discharge in exacerbations of COPD. Thorax. 2015 Dec;70(12):1123-30. doi: 10.1136/thoraxjnl-2015-207188. Epub 2015 Jul 20. PMID 26194996